CLINICAL TRIAL: NCT00460668
Title: A Prospective Single Centre Open Randomized Trial on the Effect of Post-thoracotomy Pulmonary Rehabilitation on Quality of Life
Brief Title: The Effect of Post-thoracotomy Pulmonary Rehabilitation on Quality of Life
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Isala (Other)
Responsible Party: Principal Investigator, Jan W.K. van den Berg, Dr., Isala
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: NL14089.075.06
Record Dates: First submitted 2007-04-13; First posted 2007-04-16 (Estimated); Last update posted 2013-04-08 (Estimated); Status verified 2013-04

CONDITIONS: Lung Cancer; Thoracotomy; Pulmonary Rehabilitation
Keywords: elective thoracotomy; pulmonary rehabilitation; quality of life
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Pulmonary rehabilitation post-thoracotomy (Experimental): Pulmonary rehabilitation post-thoracotomy
  Interventions: Behavioral: pulmonary rehabilitation
- Control (No Intervention): Control

INTERVENTIONS:
Behavioral: pulmonary rehabilitation — 2 or 3 times a week during 8 weeks
  Arms: Pulmonary rehabilitation post-thoracotomy

SUMMARY:
The purpose of this study is to evaluate the effects of an integrated multidisciplinary rehabilitation program on health related quality of life in the 12 months postoperative period in patients with an elective thoracotomy and to evaluate the effects of the program on general quality of life (SF-36), acute/chronic post-thoracotomy pain, impairment (changes in pulmonary function), disability (exercise capacity) and start to complete recovery (ECOG score of 0 or 1) 12 months postoperatively in patients with an elective thoracotomy.

DETAILED DESCRIPTION:
Morbidity in the post operative phase of thoracotomies is characterised by pain, dyspnea, shoulder dysfunction and a loss of exercise tolerance may occur. There is literature about post-thoracotomy painsyndromes and postoperative quality of life has been investigated. However, data on post-thoracotomy rehabilitation and influence on morbidity and recovery are not available.

Aim of the study:

Primary: To evaluate the effects of an integrated multidisciplinary rehabilitation program on health related quality of life in the 12 months postoperative period in patients with an elective thoracotomy.

Secondary: To evaluate the effects of the program on general quality of life (SF-36), acute/chronic post-thoracotomy pain, impairment (changes in pulmonary function), disability (exercise capacity) and start to complete recovery (ECOG score of 0 or 1) 12 months postoperatively in patients with an elective thoracotomy.

Study design: prospective single-centre, open randomised trial. Eighty-eight elective thoracotomy patients with an age between the 18 and 80 years will be recruited during two years. The follow up for each patient will be one year. The exclusion criteria are chronic pain involvement, a previous thoracotomy, comorbidity limiting rehabilitation, psychiatric illness and non- compliance.

Patients will be asked for participation before thoracotomy by informed consent and will be randomised post-thoracotomy, before discharge into a rehabilitation or 'regular care' group. Randomisation will take place for rehabilitation or regular care by a minimisation program with special attendance to age (< 70 or ≥ 70 years), gender, the result of the 6 minute walk test (< 100 m or ≥ 100 m), the FEV (FEV1< 40% or ≥ FEV1 40 %) and type of surgery (pneumectomy vs other). During screening a spirometry and a 6 minute walk test will be performed. The first questionnaires (VAS, McGill pain questionnaire) will be given to the patients after enrolment and before thoracotomy. The post-thoracotomy pain management consists of the standard analgetic treatment; a thoracic epidural catheter which will be slowly replaced by paracetamol, opioids and NSAID's. The consumption of analgetics will also be documented in the follow up. Supplementary oxygen and lung inhalation is given when necessary. This will be scored too. Regular physical therapy will be started directly after thoracotomy as soon as possible.

The rehabilitation program will be initiated within a month after discharge. The degree of the rehabilitation program will be separately detected for each patient by a cycle test (heart rate) within 3 weeks post-thoracotomy. Patients in the pulmonary rehabilitation program will be guided by a multidisciplinary team of pulmonologist, physical therapist and social worker during 12 weeks. The program will last 3 x 2 hours weekly consisting of exercise training and education.

All patients will be followed up after discharge at 1 month, 3 months, 6 months and 12 months at the outpatient clinic of the pulmonology department and the pain clinic of the anaesthesia department. Before discharge and at these intervals (except for the SGRQ at 1 month), patients have to fill questionnaires about quality of life (SF-36 and SGRQ) and pain (McGill pain questionnaire and VAS). Exercise capacity by means of the 6 minutes walk test and spirometry will be measured after the accomplishment of the rehabilitation program at 3 months.

During follow up all the results between the experimental rehabilitation group and the regular care group will be compared. In the interpretation of these results start to complete recovery is defined as ECOG 0 and 1.

Randomisation, blinding and treatment allocation Randomisation will take place for rehabilitation or regular care by a minimisation program with special attendance to age (< 70 or ≥ 70 years), gender, the result of the 6 minute walk test (< 100 m or ≥ 100 m), the FEV1 (FEV1< 40% or ≥ FEV1 40 %), and type of surgery (pneumectomy vs other).

Study population:

Eighty-eight patients with an elective thoracotomy between the age of 18 and 80 years.

Intervention:

An early pulmonary rehabilitation program during 12 weeks initiated after discharge from the hospital.

Inclusion criteria:

1. elective, thoracotomy patients with a surgical intention to cure.
2. age between 18 and 80 years.
3. ECOG 0 - 2 post-thoracotomy.

Exclusion criteria:

1. patients with chronic pain.
2. a previous thoracotomy.
3. comorbidity limiting rehabilitation.
4. non-compliance.

Main study endpoints

1. health related quality of life (SGRQ score). Secondary study endpoints

1. general quality of life (SF-36).
2. acute / chronic post-thoracotomy pain (McGill and VAS).
3. impairment (changes in pulmonary function).
4. disability (exercise capacity; 6 Minute Walking Distance).
5. start to complete recovery (ECOG score of 0 or 1).

Statistical analysis: All analysis will be on an intention-to-treat basis. The primary analysis will be on an intention-to-treat basis. The mean change in the primary endpoint (SGRQ total score) after 6 months between the groups will be analysed using unpaired t-tests. These tests will also be used to analyse differences after 12 months in secondary endpoints (SF-36 scores, 6-minute walking difference, pain scores, and lung function values). Since some study endpoints (quality of life and pain scores) will be measured more than two times (repeatedly measured) the course of these scores in time will be tested using MANOVA-analysis. To test for differences in proportions (proportion of patients with an ECOG-score of 0 or 1 after rehabilitation) the Chi2 -test will be used.

Burden and risks associated with participation:

There are no adverse effects due to the rehabilitation program. Patients in the 'regular care' group will not be guided by the multidisciplinary rehabilitation team. The disadvantages are the following: Patients have to fill in quality of life questionnaires, pain questionnaires and have to evaluate painscales (SGRQ, SF-36; McGill Pain questionnaire and VAS) have to perform the 6 minutes walk-test and a spirometry twice. Finally, patients have to visit the pulmonologist and the pain clinic more frequently. The expected benefits are a better exercise tolerance, less pain and a better quality of life; a faster recovery.

ELIGIBILITY:
Inclusion Criteria:

* elective, thoracotomy patients with a surgical intention to cure.
* age between 18 and 80 years.
* ECOG 0 - 2 post-thoracotomy.

Exclusion Criteria:

* patients with chronic pain.
* a previous thoracotomy.
* comorbidity limiting rehabilitation.
* non-compliance

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2007-04; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
SGRQ total score | 12 months

SECONDARY OUTCOMES:
SF-36 scores | 12 months
McGill pain questionnaire scores | 12 months
Pulmonary function and 6MWD | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: J.A. Stigt, Study Director — Isala
Locations (1):
- Isala Klinieken, Zwolle, Netherlands